CLINICAL TRIAL: NCT00001853
Title: Diabetes and Heart Disease Risk in Blacks
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990002; 99-DK-0002
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-30

CONDITIONS: Cardiovascular Diseases; Diabetes; Obesity; Hypertension
Keywords: Healthy Volunteers; Health Disparities; Diabetes; Cardiovascular Disease; Natural History
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Obesity; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy adult African Americans born in the United States, with American born parents or born in Africa with African born parents.

SUMMARY:
It is unknown if obesity contributes to the development of heart disease in African American men and women.

This study was created to determine whether there is a relationship between sex and body size and the incidence of heart disease in African American men and women. Researchers will attempt to associate obesity with the presence of heart disease risk factors. Risk factors that will be studied include; total body fat, body fat distribution, fat content of the blood (triglyceride concentration, low density lipoproteins [LDL], and high density lipoproteins [HDL]), how fast fat is removed from the blood, and how well insulin works in the body.

Scientific studies have shown that obesity and increased levels of fat content in the blood are important risk factors for heart disease in Caucasian women. However, similar studies in African American women have failed to show the same correlation. In fact, it appears that African American women in all three body weight groupings, nonobese, overweight, and obese experience high death rates due to heart disease. In addition, prior research has shown that obese African American men tend to have elevated levels of fat in the blood while African American women have normal blood fat levels. Therefore, if high levels of triglycerides (fat found in the blood) are not seen in non-diabetic obese African American women, it cannot be considered a risk factor in this population. This suggests that studies conducted on Caucasian women may not provide insight into heart disease risk factors in African American women.

The study will take 2000 healthy non-diabetic African American men and women (ages 18-70) and body mass index 3 subgroups; nonobese, overweight and obese. Diabetes undeniably increases the risk of heart disease. Therefore patients suffering from diabetes will not be included in the study. Candidates for the study will undergo a series of tests and examinations over 2 outpatient visits. Subjects will have body fat analyses, resting energy expenditure measurements, an EKG (electrocardiogram), and specific blood tests.

Researchers believe this study will provide significant insight into the causes of obesity and heart disease in African Americans.

DETAILED DESCRIPTION:
This study is designed to investigate in blacks the relationship of risk for diabetes and heart disease from obesity plasma glucose and triglyceride concentrations and the triglyceride related risk factors of small dense low density lipoprotein (LDL), high density lipoprotein (HDL) and central obesity.

The Framingham Study demonstrated that obesity and elevated glucose and triglyceride levels are important risk factors for coronary artery disease in white women. However, studies that have had significant participation of black women such as the Charleston Heart Study, failed to show a relationship of obesity or triglyceride to coronary artery disease mortality in black women. In fact, black women independent of body weight or triglyceride levels experience high mortality from coronary artery disease. Our earlier research has demonstrated that obese black men have elevated triglyceride levels but obese black women have normal triglyceride levels. Consequently if elevated triglyceride levels do not occur in obese nondiabetic black women, then elevated triglyceride levels may not represent a major cardiovascular risk for black women.

The study, Diabetes and Heart Disease Risk in Blacks, is designed to determine the role of obesity, glucose and triglyceride on risk for heart disease in blacks. For this study of blacks, we will study 2 groups, African Americans and Black Africans living in the United States. African Americans must self-identify as African American, be born in the United States and have parents who self-identify as African American and were born in the United States. The second group will be blacks living in the United States but were born in Africa and whose parents were born in Africa.

We will recruit 2000 healthy, non-diabetic individuals (), age range 18- 70, and body mass index (3 subgroups: nonobese, overweight and obese). In 2 outpatient visits to the Clinical Center, participants will have body fat analyses, an electrocardiogram, an oral glucose tolerance test, questionnaires about sleep, stress, discrimination, resilience, etc. and an intravenous glucose tolerance test or a beverage tolerance test. This study has the potential to provide significant insight and lead to the development of programs that help

decrease diabetes and cardiovascular risk in blacks.

ELIGIBILITY:
* IINCLUSION AND EXCLUSION CRITERIA

CRITERIA FOR INCLUSION:

Ethnicity: Black

This is a study of adult African Americans and Blacks that were born in Africa but are now living in the United States. As African American people are multi-ethnic, we will in this initial investigation, study two different groups of African American. To enroll participants must self-identify as African Americans and be born in the United States, with American born parents or be born in Africa with African born parents. In both groups we will study sex differences in the role of obesity and TG levels on cardiovascular disease. In the future, we plan to expand the study to include other groups which self-identify as African Americans (i.e.AfroCarribeans and Hispanic blacks).

Only blacks are included in this study because the focus of this study is on gender differences in blacks in risk factors for CAD, specifically obesity, TG levels and TG related CAD risk factors. Unlike Caucasian women, premenopausal black women do not appear to be as protected from heart disease as a result of their gender. One model to study this apparent decrease in gender

related cardioprotection in black women is to compare black men to black women. An alternative model would be to compare black women to Caucasian women. However, since the primary focus of this work is on gender differences rather than racial differences comparing black women to men is a superior model. Other racial groups do not share the loss of gender-related cardioprotection found in blacks, and have been excluded. Further the advantage of comparing black men and women is that this comparison provides a better control of dietary, cultural and genetic factors.

Age: The age range of the participants will be between 18 and 70 years. As stated in the original protocol on page 14: Future investigations are planned which will involve similar comparisons between premenopausal and postmenopausal black women and between whites and blacks. To investigate risk for glucose intolerance, diabetes and cardiovascular risk factors, it is no longer sufficient to maintain the age range between 18 and 50 years. We need to expand to an age range with an increased prevalence of these risk factors.

Medical History: To participate in the study subjects should identify themselves as healthy. This is important so the broadest possible sample of people will enroll. The fact that people are healthy will be confirmed by the history, physical and laboratory tests done as part of the screening visit. People with established coronary artery as evidenced by history of myocardial infarction, coronary artery bypass surgery or PTCA will be allowed to participate if they are not currently having angina.

CRITERIA FOR EXCLUSION:

Black Ethnicity other than American or African.

As stated in the inclusion criteria black people are a multi-ethnic group. In this initial investigation we are focusing on African Americans who are American born and Africans living in the United States who are African born. In the future, we will expand the study to include other groups of blacks such as individuals of Afro-Caribbean and Hispanic blacks.

Medications: People who take medications that are known to alter the parameters which are under investigation in this study will be excluded. People taking medications to treat hyperlipidemia will be included but analyses will be adjusted to take this into account. Subjects on thyroid hormone replacement will be included if their TSH is normal.

Diabetes: Because diabetes affects insulin sensitivity and TG levels all people with diabetes even if the diabetes is controlled with diet alone will not be enrolled in the study.

Pregnant or Breastfeeding: Women who are pregnant, breastfeeding, or have an infant that is less than four months of age will be excluded. This is because the physiologic changes associated with pregnancy, breastfeeding or recent childbirth affect the parameters under study.

Menstrual History: Now that postmenopausal women are included, menstrual history will be taken but women with irregular menses and hysterectomy will not be excluded. Women between the ages of 40 and 55 years will have FSH checked for proper characterization. Women 56 years of age and older will be assumed to be postmenopausal. However, women on any type of injectable hormonal contraception will be excluded because hormonal contraception affects both TG levels and glucose metabolism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers of African descent,specifically African-born blacks and African Americans, recruited from the local area by flyer, newspaper advertisements, word of mouth and study personnel describing the study at community events.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1998-10-21 (Actual)

PRIMARY OUTCOMES:
Diabetes and Heart Disease Risk | By Subject
  Glucose Tolerance Status Lipid Profile Sickle Cell Trait Status Glucose 6 Phosphate Dehydrogenase Activity

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Sumner, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Undetermined at this time

REFERENCES:
- [Background] Utumatwishima JN, Chung ST, Bentley AR, Udahogora M, Sumner AE. Reversing the tide - diagnosis and prevention of T2DM in populations of African descent. Nat Rev Endocrinol. 2018 Jan;14(1):45-56. doi: 10.1038/nrendo.2017.127. Epub 2017 Oct 23. PMID 29052590
- [Background] Kabakambira JD, Baker RL Jr, Briker SM, Courville AB, Mabundo LS, DuBose CW, Chung ST, Eckel RH, Sumner AE. Do current guidelines for waist circumference apply to black Africans? Prediction of insulin resistance by waist circumference among Africans living in America. BMJ Glob Health. 2018 Oct 15;3(5):e001057. doi: 10.1136/bmjgh-2018-001057. eCollection 2018. PMID 30364383
- [Background] Briker SM, Aduwo JY, Mugeni R, Horlyck-Romanovsky MF, DuBose CW, Mabundo LS, Hormenu T, Chung ST, Ha J, Sherman A, Sumner AE. A1C Underperforms as a Diagnostic Test in Africans Even in the Absence of Nutritional Deficiencies, Anemia and Hemoglobinopathies: Insight From the Africans in America Study. Front Endocrinol (Lausanne). 2019 Aug 7;10:533. doi: 10.3389/fendo.2019.00533. eCollection 2019. PMID 31447780
- [Derived] Wentzel A, Duhuze Karera MG, Patterson AC, Waldman ZC, Schenk BR, Mabundo LS, DuBose CW, Horlyck-Romanovsky MF, Sumner AE. The Africans in America study demonstrates that subclinical cardiovascular risk differs by etiology of abnormal glucose tolerance. Sci Rep. 2022 Oct 10;12(1):16947. doi: 10.1038/s41598-022-19917-8. PMID 36216842
- [Derived] Ishimwe MCS, Wentzel A, Shoup EM, Osei-Tutu NH, Hormenu T, Patterson AC, Bagheri H, DuBose CW, Mabundo LS, Ha J, Sherman A, Sumner AE. Beta-cell failure rather than insulin resistance is the major cause of abnormal glucose tolerance in Africans: insight from the Africans in America study. BMJ Open Diabetes Res Care. 2021 Sep;9(1):e002447. doi: 10.1136/bmjdrc-2021-002447. PMID 34531244
- [Derived] Jagannathan R, DuBose CW, Mabundo LS, Chung ST, Ha J, Sherman A, Bergman M, Sumner AE. The OGTT is highly reproducible in Africans for the diagnosis of diabetes: Implications for treatment and protocol design. Diabetes Res Clin Pract. 2020 Dec;170:108523. doi: 10.1016/j.diabres.2020.108523. Epub 2020 Oct 22. PMID 33153960
- [Derived] Hobabagabo AF, Osei-Tutu NH, Hormenu T, Shoup EM, DuBose CW, Mabundo LS, Ha J, Sherman A, Chung ST, Sacks DB, Sumner AE. Improved Detection of Abnormal Glucose Tolerance in Africans: The Value of Combining Hemoglobin A1c With Glycated Albumin. Diabetes Care. 2020 Oct;43(10):2607-2613. doi: 10.2337/dc20-1119. Epub 2020 Aug 14. PMID 32801129
- [Derived] Briker SM, Hormenu T, DuBose CW, Mabundo LS, Chung ST, Ha J, Sherman A, Tulloch-Reid MK, Bergman M, Sumner AE. Metabolic characteristics of Africans with normal glucose tolerance and elevated 1-hour glucose: insight from the Africans in America study. BMJ Open Diabetes Res Care. 2020 Jan;8(1):e000837. doi: 10.1136/bmjdrc-2019-000837. PMID 31958302
- [Derived] Bingham BA, Duong MT, Ricks M, Mabundo LS, Baker RL Jr, Utumatwishima JN, Udahogora M, Berrigan D, Sumner AE. The Association between Stress Measured by Allostatic Load Score and Physiologic Dysregulation in African Immigrants: The Africans in America Study. Front Public Health. 2016 Nov 25;4:265. doi: 10.3389/fpubh.2016.00265. eCollection 2016. PMID 27933289
- [Derived] Sumner AE, Duong MT, Bingham BA, Aldana PC, Ricks M, Mabundo LS, Tulloch-Reid MK, Chung ST, Sacks DB. Glycated Albumin Identifies Prediabetes Not Detected by Hemoglobin A1c: The Africans in America Study. Clin Chem. 2016 Nov;62(11):1524-1532. doi: 10.1373/clinchem.2016.261255. Epub 2016 Sep 13. PMID 27624138
- [Derived] Polidori DC, Bergman RN, Chung ST, Sumner AE. Hepatic and Extrahepatic Insulin Clearance Are Differentially Regulated: Results From a Novel Model-Based Analysis of Intravenous Glucose Tolerance Data. Diabetes. 2016 Jun;65(6):1556-64. doi: 10.2337/db15-1373. Epub 2016 Mar 18. PMID 26993071
- [Derived] Sumner AE, Duong MT, Aldana PC, Ricks M, Tulloch-Reid MK, Lozier JN, Chung ST, Sacks DB. A1C Combined With Glycated Albumin Improves Detection of Prediabetes in Africans: The Africans in America Study. Diabetes Care. 2016 Feb;39(2):271-7. doi: 10.2337/dc15-1699. Epub 2015 Dec 17. PMID 26681716
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1999-DK-0002.html